CLINICAL TRIAL: NCT05899283
Title: A Randomized, Crossover, Controlled Clinical Study of the Capillary High-Flux Hemodialysis Filters OCI-HF160 and FX800HDF
Brief Title: A Comparative Study of Two Kinds of Hemodialysis Filters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jianhui Zhou, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S2021-171-01
Record Dates: First submitted 2023-01-31; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Uremia
Keywords: Hemodialysis Filter; OCI-HF160; FX800HDF
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A(OCI-HF160+FX800HDF) (Experimental): Group A first used the hemodialysis filter OCI-HF160, then used FX800HDF.
  Interventions: Device: OCI-HF160; Device: FX800HDF
- Group B(FX800HDF+OCI-HF160) (Experimental): Group B first used the hemodialysis filter FX800HDF, and then used OCI-HF160.
  Interventions: Device: OCI-HF160; Device: FX800HDF

INTERVENTIONS:
Device: OCI-HF160 — OCI-HF160 are used in patients for hemofiltration, hemodialysis and hemodiafiltration, to correct solute and fluid imbalances in patients' blood.
  Other Names: the Chengdu Ousai Hollow Fiber Membrane Hemodialysis Filter OCI-HF160
Device: FX800HDF — FX800HDF are used in patients for hemofiltration, hemodialysis and hemodiafiltration, to correct solute and fluid imbalances in patients' blood.
  Other Names: the Fresenius Hemodialysis Filter FX80

SUMMARY:
This study exploring the expression characteristics of different cells of peripheral blood after exposure to two kinds of hemodialysis filter membrane materials will help to elucidate the key mechanisms of hemodialysis filter coagulation occurrence, which is an important guideline for reducing the occurrence of adverse events in hemodialysis.

DETAILED DESCRIPTION:
Background: Hemodialysis is one of the important alternative treatments for patients with uremia, and effective hemodialysis treatment can improve mortality and quality of life. However, during hemodialysis treatment, contact between blood and artificial materials often triggers a coagulation cascade reaction, which induces dialyzer coagulation. Studies have found that the incidence of dialyzer coagulation ranges from 5% to 14%. Once coagulation occurs, it inevitably affects the efficiency of the patient's dialysis and may lead to interruption of dialysis and blood loss, with the serious possibility of systemic thromboembolic events. To prevent clotting, systemic anticoagulation is usually required, which inevitably increases the risk of bleeding and lacks safe and effective anticoagulation methods. Some studies have suggested that the endogenous coagulation pathway is the primary pathway of dialyzer coagulation and that coagulation is effectively prevented by the use of antibodies to coagulation factor F Ⅻ during extracorporeal circulation. Some studies, however, suggest that the exogenous coagulation pathway is the primary pathway of dialyzer coagulation. An in-depth study of coagulation activation will help us to understand the true mechanism of dialyzer coagulation occurrence and provide new targets for the prevention and treatment of coagulation during dialysis.

Methods: The study population consisted of 10 patients with uremia newly placed on hemodialysis treatment for the first time. Inclusion criteria: 1.70 years ≥age ≥ 18 years, gender not limited; 2.Patients with clinical diagnosis of chronic renal insufficiency (CKD stage 5) requiring renal replacement therapy; 3.Dialysis access was central venous catheter; 4.Newly placed tubing, not dialysed patients; 5.Patients voluntarily participated and written informed consent signed by the patient or authorized delegate had been obtained.Exclusion criteria: 1.Patients with acute renal failure; 2.Patients are participating in other clinical studies; 3.Pregnancy or breastfeeding; 4.Use of hemostatic or anticoagulant drugs in the last 1 week; 5.Positive infectious serum markers for HIV, syphilis, hepatitis B, and hepatitis C; 6. Presence of active infection; 7.Allergy to dialyzers.Observation index: Peripheral blood before and after dialysis and filter after dialysis were collected, and blood routine, coagulation factors, single cell sequencing and electron microscopy were performed to compare the changes of coagulation factor activity before and after contact with dialysis membrane, and to screen the major coagulation factors and coagulation pathway activation pathways. Single-cell transcriptome characteristics of peripheral blood mononuclear cells before and after exposure to dialysis membranes were analyzed to explore the key mechanisms of peripheral blood cells regulating coagulation contact activation. Statistical methods: SPSS version 17.0 statistical software was applied for statistical analysis, and continuous variables were expressed as mean ± standard deviation, and non-continuous variables were expressed as percentages. Comparisons between two data were made by independent t-test or χ2 test, and P<0.05 was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, gender not limited;
2. Patients with clinical diagnosis of chronic renal insufficiency (CKD stage 5) requiring renal replacement therapy;
3. Dialysis access was central venous catheter;
4. Newly placed tubing, not dialysed patients; (5) patients voluntarily participated and written informed consent signed by the patient or authorized delegate had been obtained.

Exclusion Criteria:

1. Patients with acute renal failure;
2. Patients are participating in other clinical studies;
3. Pregnancy or breastfeeding;
4. Use of hemostatic or anticoagulant drugs in the last 1 week;
5. Positive infectious serum markers for HIV, syphilis, hepatitis B, and hepatitis C;
6. Presence of active infection;
7. Allergy to dialyzers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Filter coagulation grade 3 | 4 hours
  Filter coagulation grade 3 is a severe clotting events
Filter multiplexer residual volume <0.8 | 4 hours
  Filter multiplexer residual volume <0.8 is also a severe clotting events

SECONDARY OUTCOMES:
Blood platelets | 4 hours
  The normal value of blood platelets is 100×10^9/L~300×10^9/L
Hemoglobin | 4 hours
  The normal values are 120-160g/L for adult males and 110-150g/L for adult females
Leukocytes | 4 hours
  The normal value is 4×10^9/L~10×10^9/L
Blood coagulation factor TF | 4 hours
  TF is the initiating factor of coagulation reaction
Blood coagulation factor FXII | 4 hours
  Coagulation factor FXII is a protease involved in the blood coagulation pathway
Blood coagulation factor F1+2 | 4 hours
  Coagulation factor F1+2 can reflect thrombin activity
Scanning electron microscope | 4 hours
  Scanning electron microscopy to observe the area of the dialyzer fibrous clot as a percentage of the entire field of view
Single-cell transcriptome sequencing | 4 hours
  With the consent of the patients, blood were taken for analysis. Isolation of lymphocytes from blood to measure its gene expression profile
Transmembrane pressure | 4 hours
  Transmodular pressure changes were recorded every 15 minutes during dialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China